CLINICAL TRIAL: NCT00449059
Title: Acute Effect of Nitroglycerin on Cyclosporine-Induced Hypertension After Cardiac Transplantation
Brief Title: Nitrate and Hypertension in Heart Transplanted Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nitrate_USZ04
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2007-03-19 (Estimated); Status verified 2007-03

CONDITIONS: Hypertension; Heart Transplantation
Keywords: heart transplantation; cyclosporine; hypertension; nitroglycerin
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: acute infusion of nitroglycerine into the pulmonary artery

SUMMARY:
The aim of the study was to evaluate the acute effect of nitroglycerine infusion on blood pressure and heart rate in heart-transplanted patients with cyclosporine-induced hypertension.

DETAILED DESCRIPTION:
Background: Cyclosporine represents a milestone in immunosuppression after organ transplantation. Its use, however, comes at the cost of significant side effects, such as arterial hypertension. Our aim was to investigate the effect of acute administration of nitroglycerin in heart-transplanted patients with cyclosporine-induced hypertension.

Methods: We included 18 hypertensive patients (HT) scheduled for elective cardiac catheterization after heart transplantation and treated with cyclosporine, as well as 6-matched HT. Simultaneous measurements of BP in the aorta and pulmonary artery before and after administration of nitroglycerin were done.

Results: After injection of 50μg and 100μg nitroglycerin a significant BP decrease was observed both in heart-transplanted patients (sBP p=0.0001; dBP p=0.0001) and in controls (sBP p=0.006; dBP p=0.05). This reduction was more pronounced in heart-transplanted patients (sBP p=0.022; dBP 0.018 for group comparison). 8±3 minutes after the last nitrate infusion BP remained significantly reduced vs baseline in heart-transplanted patients (p<0.001) while it comes back to baseline in controls. The reduction in sBP (p=0.04 after 50μg nitroglycerin; p=0.05 after 100μg nitroglycerin) but not dBP correlated to cyclosporinemia.

Conclusions: This study indicates that nitroglycerin reduces sBP in heart-transplanted patients with cyclosporine-induced hypertension. Further studies are needed to evaluate the long-term effect of nitrates in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Heart-transplanted group:
* Patients with hypertension and treated with cyclosporine
* Patients under optimal standard therapy
* Patients giving written informed consent

Control group:

* Patients with hypertension
* Patients without prior transplantation of any kind
* Patients giving written informed consent

Exclusion criteria:

* Hypertensive patients receiving immunosuppressive drugs
* Patients receiving any kind or nitrate derivates

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-01; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure reduction after acute nitroglycerine infusion

SECONDARY OUTCOMES:
Heart rate modification after acute nitroglycerine infusion

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Corti, MD, Principal Investigator — Cardiovascular Center, University Hospital Zurich, Zurich, Switzerland
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland